CLINICAL TRIAL: NCT04353102
Title: A First-in-Human (FIH), Multicenter, Open-Label, Phase 1 Dose-Escalation Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of YH002 in Subjects With Advanced Solid Malignancies
Brief Title: A Study to Evaluate the Safety, Tolerability and How YH002 Enters, Moves Through and Exits the Body in Subjects With Advanced Solid Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eucure (Beijing) Biopharma Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: YH002002
Record Dates: First submitted 2020-04-17; First posted 2020-04-20 (Actual); Last update posted 2022-07-22 (Actual); Status verified 2022-07

CONDITIONS: Advanced Solid Malignancies
Keywords: dose escalation; safety; tolerability; advanced solid malignancie; pharmacokinetics

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- YH002 (Experimental): All subject will receive YH002 intravenously as single agent every three weeks (Q3W) for up to 2 years, until intolerable toxicity, confirmed disease progression, withdrawal of consent, or Investigator decision, whichever comes first. Subjects who remain on treatment in the absence of disease progression for more than 2 years may continue to receive study drug through a single patient IND.
  Interventions: Drug: YH002

INTERVENTIONS:
Drug: YH002 — YH002 will be administered intravenously every three weeks (Q3W) for up to 2 years at doses of Dose A, Dose B, Dose C, Dose D, Dose E, Dose F, Dose G, and Dose H.

SUMMARY:
This is an open-label, dose-escalation study of the study drug YH002. The study is designed to determine the safety, tolerability and maximum tolerated dose (MTD) and recommended Phase 2 dose (RP2D) of YH002 in patients with advanced solid Malignancies

DETAILED DESCRIPTION:
This is a single arm clinical trial in subjects with advanced solid tumor receiving multiple doses of YH002 intravenously (IV). YH002 will be administered (IV) in 6-48 patients with advanced solid tumors. An accelerated titration method followed by a traditional 3+3 dose escalation algorithm will be utilized to determine MTD/MAD. Patients will be dosed at Dose A, Dose B, Dose C, Dose D, Dose E, Dose F, Dose G, and Dose H every 3 weeks (Q3W).

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged ≥ 18 years
* Confirmed as histologically or cytologically, locally advanced or metastatic non-resectable solid tumors, must have received and progressed on, or been ineligible for, or intolerant of available standard therapies known to confer clinical benefit or for whom no standard therapy exits
* Subjects enrolled in Dose D, Dose E, Dose F, Dose G, and Dose H cohorts must have at least one measurable lesion per RECIST v1.1
* Eastern Cooperative Oncology Group (ECOG) performance status score 0 or 1 and life expectancy no less than 3 months
* Recovery, to Grade 0-1, from adverse events related to prior anticancer therapy except alopecia, < Grade 2 sensory neuropathy, lymphopenia, and endocrinopathies controlled with hormone replacement therapy

Exclusion Criteria:

* Symptomatic central nervous system (CNS) metastases. Subjects with asymptomatic CNS metastases who are radiologically and neurologically stable ≥ 4 weeks following CNS- directed therapy, and do not require corticosteroids or anticonvulsants are eligible for study entry
* Received anticancer therapy or radiation therapy within 5 half-lives or 4 weeks prior to study entry, whichever is shorter
* Received palliative radiotherapy to a single area of metastasis within 2 weeks prior to study entry
* Received agonist antibodies to TNFR such as anti-CD137, OX40, CD27 and CD357 antibodies prior to the study entry
* Allergy or sensitivity to YH002, or known allergies to antibodies produced from Chinese hamster ovary cells which assessed to increase the potential for an adverse hypersensitivity to YH002 by Investigator
* History of a Grade 3-4 allergic reaction to treatment with another monoclonal antibody
* Grade ≥3 irAEs or irAEs that lead to discontinuation of prior immunotherapy. Hypothyroidism, Type 1 DM, and dermatologic irAEs (except previous Steven Johnson Syndrome, toxic epidermal necrolysis, or other severe forms of dermatitis). Type 1 DM should be controlled with reduction of toxicity to Grade 1 or less
* Concomitant active autoimmune disease or history of autoimmune disease requiring systemic treatment or history of autoimmune disease within 2 years prior to study entry (except vitiligo, resolved childhood asthma/atopy, type I diabetes mellitus or hypothyroidism which can be managed by replacement therapy)
* Received steroids or other immunosuppressive systemic therapy within 4 weeks prior to the first dose of the study drug, or has need to be treated during the study (except using on low systemic absorption location prevent or treat non- autoimmune condition)
* Active hepatitis B or C. Hepatitis B carriers without active disease or cured Hepatitis C may be enrolled
* Severe cardiovascular disease within 6 months of study entry

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2020-04-22 (Actual); Primary Completion 2021-09-14 (Actual); Study Completion 2021-11-24 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events and serious adverse events | From screening up to 2 year
  The safety profile of YH002 will be assessed by monitoring the adverse events (AE) per the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) v5.0
Maximum tolerated dose (MTD) | Cycle 1 of each cohort. Duration of one cycle is 3 weeks
  MTD is defined as the highest dose level at which no more than 1 out of 6 subjects experiences a DLT during the first cycle
Dose-limiting toxicities (DLT) | Cycle 1 of each cohort. Duration of one cycle is 3 weeks
  DLT is defined as a toxicity (adverse event at least possibly related to YH002) occurring during the DLT observation period (the initial 21 days)

SECONDARY OUTCOMES:
Area under the serum concentration versus time curve within one dosing interval (AUCtau) | Up to 2 years
  To determine the pharmacokinetics (PK) profile of YH002
Volume of distribution (Vd) | Up to 2 years
  To determine the pharmacokinetics (PK) profile of YH002
Volume of distribution at steady state (Vss) | Up to 2 years
  To determine the pharmacokinetics (PK) profile of YH002
Maximum serum concentration (Cmax) | Up to 2 years
  To determine the PK profile of YH002 as single agent
Trough concentration before the next dose is administered (Ctrough) | Up to 2 years
  To determine the PK profile of YH002
Time to reach maximum serum concentration (Tmax) | Up to 2 years
  To determine the PK profile of YH002
Clearance (CL) | Up to 2 years
  To determine the PK profile of YH002
Terminal half-life (T1/2) | Up to 2 years
  To determine the PK profile of YH002
Dose proportionality | Up to 2 years
  To determine the PK profile of YH002
Incidence of anti-drug antibodies (ADAs) | Up to 2 years
  To assess the immunogenicity of YH002
Incidence of neutralizing antibodies (NAbs) | Up to 2 years
  To assess the immunogenicity of YH002
Objective response rate (ORR) | Up to 2 years
  To assess the preliminary antitumor activity of YH002
Duration of response (DOR) | Up to 2 years
  To assess the preliminary antitumor activity of YH002
Progression free survival (PFS) | Up to 2 years
  To assess the preliminary antitumor activity of YH002
Time to response (TTR) | Up to 2 years
  To assess the preliminary antitumor activity of YH002
Disease control rate (DCR) | Up to 2 years
  To assess the preliminary antitumor activity of YH002
Duration of disease control (DOC) | Up to 2 years
  To assess the preliminary antitumor activity of YH002

CONTACTS AND LOCATIONS:
Locations (3):
- Australia (3):
  - St George Private Hospital, Kogarah, New South Wales
  - Macquarie University, Macquarie, New South Wales
  - Peninsula & South Eastern Haematology and Oncology Group, Frankston, Victoria